CLINICAL TRIAL: NCT02706652
Title: Prospective Screening for Patient Specific Genotypes and Phenotypes That Influence Drug Dosing and Trial Selection in Cancer Patients
Brief Title: Prospective Screening for Patient-Specific Genotypes and Phenotypes That Influence Drug Dosing and Trial Selection in Cancer Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160076; 16-C-0076
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-05-15

CONDITIONS: Cancer
Keywords: Screening; Genotype; Drug Dosing; Trial Selection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all patients: all eligible patients

SUMMARY:
Background:

People's genetic markers and other genetic characteristics can affect their response to drug therapy. Researchers want to screen people for these markers and characteristics. They want to do this before the people are screened for studies at the National Cancer Institute. That should save time that can be lost when people go through the whole screening for a study only to find out they cannot join. The data collected may also be used to select the proper dose of anticancer agents that are being studied.

Objective:

To screen people for genetic markers and/or baseline characteristics. These will be used to determine if they can enroll in a clinical trial. They may also be used to select the proper dose of anticancer agents that are being tested.

Eligibility:

Adults 18 and older who are being considered for or being treated in a National Cancer Institute study

Design:

Participants will have their blood drawn for genetic tests.

Some participants will have a cheek swab.

Participants genetic data will be stored for future research. It could be shared with other researchers.

DETAILED DESCRIPTION:
Background:

Genetic sequence of drug-metabolizing enzymes, transporters/receptors, transcription factors, drug targets, and patient baseline characteristics often affect an individual s response to drug therapy. Expression of such genes is also influenced by the epigenome and regulation by a variety of other factors: RNA expression, protein expression, disease state, comorbidities, concomitant therapies, etc. Therefore, inter-patient variability in drug pharmacokinetics and outcome is often a function of these factors.

Inter-individual differences in efficacy and toxicity of cancer chemotherapy are especially important given the narrow therapeutic index of these drugs.

During analysis of investigational agents, inter-individual variability in pharmacokinetics, pharmacodynamics, clinical outcome, and toxicity are often noted. Many of these differences are potentially clinically actionable and depend on the aforementioned markers.

Objectives:

To screen patients for genomic markers, epigenomic markers, RNA markers, protein markers, and/or baseline characteristics that are used inform either enrollment in therapeutic clinical trials or dose selection of investigational anticancer agents.

Eligibility:

All individuals seeking enrollment on National Cancer Institute clinical trials that include a priori assessment of a patients genome, epigenome, proteome, or baseline characteristics as eligibility criteria for enrollment or dose selection.

Design:

This study will be used as a screening protocol to enroll patients for a priori screening that is necessary for inclusion in IRB-approved clinical trials taking place at the NCI.

As the rationale for ascertaining the status of a marker prior to study inclusion will be presented in the associated clinical trial, the present study will be amended on a case-by-case basis.

The accrual ceiling for this study is 900 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any patient who is being evaluated for and/or treated on an IRB-approved protocol at the National Cancer Institute.
* Age >18 years.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

- A patient will be excluded if there is an insufficient quality or quantity of sample available to perform the assay and no further sample can be drawn in order to re-assess the status of a genetic or biomarker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is being evaluated for and/or treated on one of the following IRB-approved protocols at the National Cancer Institute: 12-C-0151, or 09-C-0173, or 18-C-0061.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To provide pharmacogenomic and/or biomarker analysis to support enrollment of patients on clinical trials that require such markers prior to enrollment. | duration of study
  Collection of 6 mL of peripheral blood to analyzed via DMET Plus kit for pathway genotype of enzymes and transporters with putative relevance for the drug of interest.

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0076.html